CLINICAL TRIAL: NCT05862311
Title: The Effect of Non-Surgical Periodontal Therapy on Sclerostin, Irisin, RANKL \ OPG, IL-6 and TNF-α Levels in Type 2 Diabetes and Systemically Healthy Individuals
Brief Title: The Effect of Non-Surgical Periodontal Treatment on Bone Metabolism in Type 2 Diabetes and Systemically Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Ummuhan Tekin Atay, principal investigator, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ummuhantekinatay.
Record Dates: First submitted 2023-04-16; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Periodontal Diseases
Keywords: Gingival Crevicular Fluid; Irisin; Periodontitis; Sclerostin
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Sclerosteosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systemically healthy and periodontitis (Experimental)
  Interventions: Diagnostic Test: ELISA
- type 2 diabetes and periodontitis (Experimental)
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — ELISA(enzyme-linked immunosorbent assay)

SUMMARY:
In this study, it was concluded that sclerostin and irisin may be alternative markers for evaluating the effectiveness of periodontal treatment and healing of periodontal tissues by affecting bone metabolism.

DETAILED DESCRIPTION:
Background: Diabetes and periodontitis are chronic inflammatory diseases with similar pathogenesis and clinical and immunological interrelationships. The aim of this study is to determine periodontal clinical parameters and sclerostin, irisin, Receptor Activator of Nuclear Factor κB Ligand (RANKL)/Osteoprotegerin (OPG), interleukin-6 (IL-6) and tumor necrosis factor-α (TNF-α) levels in gingival crevicular fluid (GCF) in individuals with type 2 diabetes and systemically healthy periodontitis and to evaluate the effect of non-surgical periodontal therapy on these clinical parameters and biomarkers.

Method: Within the scope of this study, applying to Necmettin Erbakan University Faculty of Dentistry Periodontology Clinic; A total of 50 individuals, including 25 patients with type 2 diabetes and periodontitis (DMP group) and 25 patients with systemically healthy and periodontitis (SSP group), were included in the study. After recording the clinical periodontal parameters (gingival index (GI), plaque index (PI), probing pocket depth (PPD), clinical attachment level (CAL)) of each individual included in the study, GCF samples were obtained and non-surgical periodontal therapy were completed. The individuals were invited to the controls 3 months later and the procedures for clinical periodontal measurements and DOS samples collection were repeated. Levels of biomarkers in DOS samples were determined by ELISA (Enzyme Linked Immunosorbent Assay) method.

ELIGIBILITY:
Inclusion Criteria:

* Having at least 20 teeth in the mouth, excluding the third molars,
* Individuals between the ages of 18-65
* Diagnosed as stage 2 or stage 3 periodontitis as a result of periodontal examination
* Those who do not have predisposing factors (restoration, caries, etc.)

Exclusion Criteria:

* Smoking or using alcohol,
* Any periodontal treatment performed in the last 6 months,
* Being in pregnancy and/or lactation period,
* Individuals who had received any anti-inflammatory, antibiotic, antioxidant or corticosteroid treatment in the last 6 months and refused to participate in the study were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of bone metabolism biomarkers in different periodontal conditions | baseline
  The levels of bone metabolism markers (such as sclerostin, irisin, IL-6, TNF-a, RANKL/OPG) in the gingival crevicular fluid of individuals with different periodontal conditions were compared using the ELISA (Enzyme Linked İmmünosorbent Assay) test, and the relationship of these markers with periodontal status was examined.

SECONDARY OUTCOMES:
Probing pocket depth | baseline
  Probing pocket depth(PPD) was measured for determining the severity of the disease and clinical outcome. High probing depth shows more severe periodontal disease.
gingival index | baseline
  The differences in gingival index scores between periodontally healthy and periodontitis.The gingival index was recorded for determining and classifying gingival status. The gingival index (Gİ) scores each site on a 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling and spontaneous bleeding.
Plaque index | baseline
  The differences in plaque index scores between periodontally healthy and periodontitis. Plaque index (PI) was recorded for determining and classifying oral hygiene status. The plaque index (PI) scores each site on a with 0 being no plaque in gingival area and 3 abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No